CLINICAL TRIAL: NCT06724965
Title: Trans STAIR: Implementing an Evidence Based Trauma Treatment With Community Led PrEP Navigation for Transgender and Nonbinary Persons Affected by Violence
Brief Title: Trans STAIR: Implementing an Evidence Based Trauma Treatment With Community Led PrEP Navigation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: Los Angeles LGBT Center (Other); RAND (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HS-2024-0209; R34MH138228 (NIH)
Record Dates: First submitted 2024-12-06; First posted 2024-12-09 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: PrEP Uptake Experiences; PrEP Adherence Experiences; Mental Health Symptoms
Keywords: PrEP; HIV prevention; Trauma; Mental Health; PrEP adherence; PrEP uptake; STAIR; Skills Training in Affect and Interpersonal Regulation; Trauma Treatment
MeSH Terms: conditions — Wounds and Injuries; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PrEP Well + Trans STAIR (Experimental): Participants assigned to this condition will be enrolled in 3 sessions of PrEP Well + 8 sessions of Trans STAIR over 90 days. PrEP Well is a multi-level implementation strategy for providing PrEP in TGD-serving contexts by integrating peer-led PrEP navigation with programming that addresses other social and structural needs of the TGD community (e.g., housing, legal, employment, gender-affirmation, primary care). Trans STAIR (Experimental Treatment) Skills Training in Affect and Interpersonal Regulation (STAIR) adapted for TGD is 8-session, group delivery of transdiagnostic evidenced-based treatment for individuals who have experienced multiple traumas. STAIR is based in cognitive-behavioral principles and delivered in a flexible manner, with demonstrated efficacy for the treatment of PTSD, depression and other mental health symptoms known to be associated with poor medication adherence.
  Interventions: Behavioral: Trans STAIR; Behavioral: PrEP Well
- PrEP Well (Active Comparator): Participants assigned to this condition will be enrolled in 3 sessions of PrEP Well over 90 days, PrEP Well is a multi-level implementation strategy for providing PrEP in TGD-serving contexts by integrating peer-led PrEP navigation with programming that addresses other social and structural needs of the TGD community (e.g., housing, legal, employment, gender-affirmation, primary care).
  Interventions: Behavioral: PrEP Well

INTERVENTIONS:
Behavioral: Trans STAIR — Skills Training in Affect and Interpersonal Regulation (STAIR) is a transdiagnostic evidenced-based mental health treatment for individuals who have experienced multiple traumas. STAIR is based in cognitive-behavioral principles and delivered in a flexible manner over 8 group sessions, with demonstrated efficacy for the treatment of PTSD and other mental health symptoms. This trial will adapt and pilot test the STAIR intervention to be culturally appropriate and acceptable for TGD persons, adding content related to TGD health and wellness, coping with minority stress, responding to stigma and microaggressions, social support, and community connectedness, self-compassion, celebrating trans joy, trans advocacy, sexual health and PrEP use.
  Arms: PrEP Well + Trans STAIR
Behavioral: PrEP Well — This pilot trial will leverage "PrEP Well," a multi-level implementation strategy for providing PrEP in TGD-serving contexts by integrating peer-led PrEP navigation with programming that addresses other social and structural needs of the TGD community (e.g., housing, legal, employment, gender-affirmation, primary care)

SUMMARY:
This pilot trial will leverage "PrEP Well," an ongoing multi-level implementation strategy for providing PrEP in transgender/gender diverse (TGD)-serving contexts by integrating peer-led PrEP navigation with programming that addresses other social and structural needs of the TGD community (e.g., housing, legal, employment, gender-affirmation, primary care). PrEP Well has been implemented at the Trans Wellness Center (TWC) in LA since 2021. TWC is a first-of-its-kind community-led, trans-affirming, TGD community center made up of 5 community-based TGD service organizations that serve the local racially and ethnically diverse TGD community. Together with our community and implementation partners this NIMH-funded R34 will adapt evidence-based Skills Training in Affect and Interpersonal Regulation (STAIR) into a trans-affirming, culturally appropriate trauma treatment for TGD persons affected by HIV and violence (Trans STAIR); evaluate the acceptability, appropriateness, and feasibility of the Trans STAIR intervention (Phase 1 beta test; Aim 1); and conduct a Type 1: Hybrid Effectiveness-Implementation pilot randomized controlled trail (Phase 2 pilot RCT; Aims 2 and 3) of PrEP Well + Trans STAIR vs. PrEP Well alone to provide preliminary support for a fully powered larger multisite R01 to test the efficacy of PrEP Well + Trans STAIR.

DETAILED DESCRIPTION:
In Phase 1, together with community and implementation partners, the investigators will adapt evidence-based STAIR into a trans-affirming, culturally appropriate trauma treatment for TGD persons affected by HIV and violence (Trans STAIR), making suggested changes and reaching consensus at each step among the team. The investigators will then evaluate the acceptability, appropriateness, and feasibility of the Trans STAIR intervention by running a preliminary test of Trans STAIR with 20 PrEP Well participants with demonstrated suboptimal PrEP adherence. The investigators will then conduct and analyze interviews with participants and staff to obtain feedback and work with our community and implementation partners to make suggested changes until the investigators reach consensus again among the team. The investigators will then conduct interviews with key leaders, administrators, and TWC staff to assess the perceived barriers to integration of Trans STAIR into the PrEP Well implementation strategy. The investigators will then select implementation strategies that will address the identified barriers. In Phase 2, the investigators will conduct a Type 1, hybrid effectiveness-implementation pilot RCT of 70 participants randomized to receive PrEP Well + Trans STAIR vs. PrEP Well alone. The overarching goals of the pilot RCT are twofold: 1) establish the feasibility, acceptability, adoptability; preliminary effects; and cost and sustainability, and potential scalability of the PrEP Well + Trans STAIR implementation intervention; and 2) estimate the non-response rates after second-stage randomization. The aims follow the phases of the EPIS (Exploration Preparation Implementation Sustainment) framework integrated with the RE-AIM (Reach, Effectiveness, Adoption, Implementation, Maintenance) framework to assess outcomes. The investigators will systematically collect important data on factors relevant to implementation during the pilot RCT, including cost data (e.g., program budgets, interview questions leadership staff) on the resources necessary to successfully deliver the PrEP Well + Trans STAIR interventions. Consistent with a Hybrid Type I design, the investigators will leverage mixed methods data from the pilot RCT in key informant interviews with 30 participants and 10 key stakeholders/staff to document the perceptions of providers regarding implementation of PrEP Well + Trans STAIR in real-world clinical settings will set the stage for a planned multisite fully powered hybrid RCT.

ELIGIBILITY:
Inclusion Criteria:

* identify as transgender or nonbinary (non-cisgender)
* be age 18 or older
* confirmed HIV-negative status
* eligible for PrEP based on CDC guidelines
* indication of clinically significant PTSD or depressive symptoms
* ability to speak and read in English and/or Spanish

Exclusion Criteria:

* under 18 years old
* cognitively impaired to the extent that it limits ability to consent
* currently in a relationship or home where violence is occurring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — transgender male, transgender female, nonbinary identity.
Enrollment: 90 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
PrEP Uptake | Collected at 30-day and at 90-day visits.
  PrEP uptake measured via SureQuick test, a rapid point-of-care diagnostic assay used to detect the presence of tenofovir diphosphate (TFV-DP) in urine.
PrEP Adherence | Collected at 90-day follow up visit
  PrEP Adherence will be assessed via Dried Blood Spot (DBS) test, a laboratory method used for the quantitative assessment of long-term levels of Tenofovir Diphosphate (TFV-DP) in the blood, helping to monitor and confirm adherence PrEP medications such as Descovy® or Truvada®. DBS levels consistent with 4 or more average doses/week were considered adherent.

SECONDARY OUTCOMES:
Depressive symptoms (PHQ-9) | Baseline, 30-day, and 90-day visits
  The PHQ-9 (Patient Health Questionnaire-9) is a self-administered screening tool designed to assess the presence and severity of depressive symptoms in individuals. It consists of nine questions that align with the diagnostic criteria for major depressive disorder, asking respondents about their feelings and behaviors over the previous two weeks. Each question is scored on a scale from 0 (not at all) to 3 (nearly every day), resulting in a total score that can range from 0 to 27. Higher scores indicate greater severity of depression, making the PHQ-9 a valuable measure for both clinical assessments and research studies aimed at evaluating treatment outcomes and mental health interventions.
Anxiety symptoms (GAD-7) | Baseline, 30-day, and 90-day visits
  The GAD-7 (Generalized Anxiety Disorder-7) is a widely recognized self-report questionnaire used to assess the severity of generalized anxiety disorder and other anxiety-related conditions. Comprising seven questions, the GAD-7 prompts respondents to evaluate how often they have experienced specific anxiety symptoms over the past two weeks, using a scale from 0 (not at all) to 3 (nearly every day). The total score ranges from 0 to 21, with higher scores indicating more severe anxiety symptoms. This measure is frequently employed in both clinical and research settings to help identify individuals experiencing significant anxiety and to monitor changes in symptoms over time, facilitating effective treatment and intervention strategies.
PTSD symptoms (PC-PTSD-5) | Baseline, 30-day, and 90-day visits
  The PC-PTSD-5 (Primary Care Post-Traumatic Stress Disorder Screen for DSM-5) is a brief, validated screening tool designed to identify individuals at risk for post-traumatic stress disorder (PTSD) based on the diagnostic criteria specified in the DSM-5. It consists of five questions that focus on the presence of key PTSD symptoms, including intrusive thoughts, avoidance behaviors, negative changes in mood and cognition, and hyperarousal, experienced in the context of a traumatic event. Respondents answer each question with one of two options: "Yes" or "No," allowing for a quick assessment of PTSD risk. The PC-PTSD-5 is particularly useful in primary care and other clinical settings for early detection and referral for further evaluation and treatment of PTSD while being user-friendly for both patients and healthcare providers.
DSM-5 Self-Rated Level 1 Cross-Cutting Symptom Measure--Adult | Baseline, 30-day, and 90-day visits
  The DSM-5 Cross-Cutting Symptoms Measurement is a comprehensive assessment tool designed to evaluate a range of mental health symptoms that may be present across various psychiatric disorders. This assessment includes 23 symptom domains, such as anxiety, depression, psychosis, and somatic symptoms, allowing clinicians to identify and assess the severity of symptoms that might not fit neatly into specific diagnostic categories. Each item on the measure is rated on a 5-point scale (0=none or not at all; 1=slight or rare, less than a day or two; 2=mild or several days; 3=moderate or more than half the days; and 4=severe or nearBy capturing cross-cutting symptoms, this tool promotes a more holistic understanding of an individual's mental health and can facilitate better treatment planning and intervention strategies. It is particularly useful in clinical settings where comorbidity is common, as it aids in identifying overlapping symptoms that may impact overall functioning and well-being.
Inventory of Interpersonal Problems (IIP-32) | Baseline, 30-day, and 90-day visits
  The Inventory of Interpersonal Problems (IIP) is a 32-item psychological assessment tool designed to evaluate interpersonal difficulties and their impact on an individual's relationships and social functioning. The IIP consists of a series of items that assess different dimensions of interpersonal problems, such as assertiveness, reliance on others, and ability to communicate effectively. Respondents indicate the degree to which they experience difficulties in various social situations, helping to identify patterns of interpersonal behavior that may contribute to distress or dysfunction. Scores range from 0-128 with higher scores corresponding with greater interpersonal levels of dysfunction. This inventory is useful in both clinical and research settings, providing insights that can guide therapeutic interventions and enhance understanding of the relational challenges individuals face, ultimately fostering improved interpersonal dynamics and personal growth.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Storholm, PhD, Principal Investigator — San Diego State University
Locations (1):
- Los Angeles LGBT Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
NIMH requires data that involve human subjects to be shared using the NDA. Quantitative data from this pilot trial will be preserved to enable sharing via NDA data of sufficient quality to validate and replicate research findings described in the DSMP. All data collected from the randomized pilot intervention trial with 70 adult participants will be shared. De-identified survey and biomedical data will be stored within the NDA secure database. A linking file with an anonymized linking variable will also be stored if multiple datasets are required. In addition, interview protocols, codebooks, deidentified coded text, and summary findings collected from TGD participants, trans community center staff, intervention providers, and leadership will be stored in the NDA database as well.
Supporting Information: Study Protocol, SAP
Time Frame: All quantitative data will be deposited to NDA 12 months after the award begins (or following the start of the pilot trial) and every six months following the usual NDA data submission dates. The research community will have access to data when the award ends. As required by the NDA, studies will also be created that contain the data used for every publication. Data associated with each publication will be made available at the time of publication. NDA studies have digital object identifiers (DOI) to aid in findability. We will include that DOI in relevant publications. NDA will make decisions about how long to preserve the data but no data have been removed or archived to date.
Access Criteria: IPD will be available to researchers, healthcare professionals, and the general public, depending on the specific policies of the sponsoring organization or regulatory requirements.